CLINICAL TRIAL: NCT01812850
Title: Effects of the Continuous Wear of Invisalign® Trays on the Temporomandibular Joints and Orofacial Muscular Complex
Status: Completed | Type: Observational
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Andrée Montpetit, Assistant professor, Doctor of Dental Medecine, Université de Montréal
Other Study IDs: 13-024-CERES-D
Record Dates: First submitted 2013-03-13; First posted 2013-03-18 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Bruxism
Keywords: Temporomandibular joint; Orofacial muscular complex; Bruxism; Clenching; Orthodontic treatment; Invisalign®
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Invisalign®: All subjects in the study (estimation of 40 subjects) will be treated using the Invisalign® appliance.

SUMMARY:
The purpose of this study is to assess temporomandibular joint (TMJ) symptoms and night muscle activity in an objective manner, in addition to daytime bruxism and clenching, as reported by the patient, following the start of orthodontic treatment with Invisalign®. A baseline evaluation of all measures will be used as control data, while different time points will be used to evaluate the evolution of patients' symptoms over the course of six months (the duration of the study).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effects of orthodontic treatment using Invisalign® on the temporomandibular joint (TMJ) and orofacial muscular complex, on the recorded number of bruxism/clenching events during sleep, and on the reported amount of bruxism/clenching events during the day.

Principal objective:

* Evaluation of the effect of continuous wear of Invisalign® trays on the TMJ and muscles of the orofacial complex.

Secondary objectives:

* Objective evaluation of the effect of Invisalign® trays on bruxism/clenching events at night.
* Subjective evaluation of the effect of Invisalign® trays on bruxism/clenching during the day.
* Evaluation of the evolution of symptoms over the course of six months.

Appointment 1:

-Initial Exam (Initial complete orthodontic record)

Appointment 2 (T0):

* Presentation of the treatment plan
* Informed consent
* iTero Scan for Invisalign
* TMJ exam (baseline)
* Diagnostic bruxism/clenching questionnaire (baseline)
* Give Electromyogram (EMG) machine to patient for night study at home (baseline)
* Instructions on how to use the EMG machine
* NB: Patient returns EMG by courier

Appointment 3:

* Delivery of Invisalign® trays #1
* Instructions on wearing the Invisalign® trays
* Take mailing information to send EMG machine by courier (EMG recording the night before Appointment 4 / T1)

Appointment 4 (T1: 2 weeks after appointment 3):

* Patient brings back EMG machine
* TMJ exam
* Daytime bruxism/clenching questionnaire
* Bonding attachments onto teeth
* Give Invisalign® trays #2
* NB: Patient will be followed every 6-8 weeks

Appointment 5 (T2: 6 months after appointment 4):

* TMJ exam
* Daytime bruxism/clenching
* Give EMG machine for night study at home
* Patient returns EMG by courier

All subjects in the study will be treated using the Invisalign® appliance. To obtain statistically and clinically significant results, it was calculated that at least 30 patients will need to complete the study. Our objective is to recruit about 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition
* No congenially permanent teeth missing (with the exception of 3rd molars)
* Patient requiring a non-extraction orthodontic treatment
* Patient followed by the University of Montreal port-graduate orthodontic clinic
* Cl.I skeletal relation (or mild cl.II / mild cl.III)
* Patient can speak and read french
* In good health
* Patient and parents accept and sign informed consent form.
* Periodontal health permits orthodontic treatment
* Adequate oral hygiene

Exclusion Criteria:

* Diagnosed TMJ's dysfunction
* Severe TMJ's dysfunction
* Lack of attendance

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients are recruited from the Department of Orthodontics of the University of Montreal
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Effects of the continuous wear of Invisalign® trays on the temporomandibular joints and orofacial muscular complex | 6 months
  RDC/TMD Research Diagnostic Criteria Method

SECONDARY OUTCOMES:
Effects of the continuous wear of Invisalign® trays on the number of bruxism/clenching events during sleep | 6 months
  Evaluation of bruxism and clenching at night with electromyogram (EMG) recordings
Effects of the continuous wear of Invisalign® trays on the reported amount of bruxism/clenching during the day | 6 months
  Bruxism and clenching questionnaire developed by Dr Gilles Lavigne (1996)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brien, DMD, Principal Investigator; Andrée Montpetit, DMD, MSc, Study Director; Nelly Huynh, PhD, Study Director
Locations (1):
- Department of Orthodontics of the University of Montreal, Montreal, Quebec, Canada